CLINICAL TRIAL: NCT01230567
Title: Comparison Between the Histological and Clinical Diagnosis of Non Healing Wounds
Status: Completed | Type: Observational
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Yaron Har-Shai, head of plastic surgery department, Carmel Medical Center
Other Study IDs: CMC-10-0032 CTIL
Record Dates: First submitted 2010-10-28; First posted 2010-10-29 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Wounds and Injuries
Keywords: Problem wounds; Non healing wounds; BCC; SCC; Vasculitis
MeSH Terms: conditions — Wounds and Injuries; Vasculitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
50 patients with non healing wounds will undergo biopsy to conclude wether there is an occult etiology for the wound.

DETAILED DESCRIPTION:
25 patients suffering from non healing wounds which have non typical features for the clinical diagnosis (such as pale granulation, raised lesions and more) will undergo biopsy of the wound.

Another 25 patients suffering from non healing wounds with typical features for the clinical diagnosis will undergo biopsy of the wound.

The hypothesis is that non healing wounds harbor undiagnosed etiologic factors such as BCC, SCC, vasculitis etc. and that some clinical features should raise our suspicion for these occult etiologies.

ELIGIBILITY:
Inclusion Criteria:

* patients with non-healing wounds (for > 6 weeks)
* consent to be included in the study
* age 18-85

Exclusion Criteria:

* patients taking anti coagulant therapy
* patients taking steroids or immunosuppressive therapy
* pregnancy
* pace maker

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from non healing wounds, which do not respond well to six weeks of adequate treatment.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
HISTOLOGY RESULTS | 04/2013
  HISTOLOGY RESULTS OF ALL WOUND BIOPSIES WILL BE COLLECTED TO ASSESS THE ACCULT ETIOLOGY RATE IN NON HEALING WOUNDS.

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Har-Shai, Prof, Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel